CLINICAL TRIAL: NCT01333345
Title: Post-Implant Performance of the EC-3 IOL ADDENDUM TO THE PROTOCOL: Clinical Evaluation of the EC-3 Hydrophobic Acrylic Posterior Chamber Aphakic Intraocular Lens
Brief Title: Post-Implant Performance of the EC-3 IOL
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Aaren Scientific Inc. (Industry)
Responsible Party: Robert Sheehan, VP of Regulatory Affairs & Quality Systems, Aaren Scientific Inc.
Other Study IDs: DC-036 Addendum
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Cataract
Keywords: Cataract replacement surgery; implantation; EC-3 IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to obtain data on the performance of the EC-3 lens at an interval of two years (and beyond) from subjects who were implanted. The primary aim of the study will be to evaluate the presence, if any, of PCO, lens glistening, and other anomalies in the subjects.

DETAILED DESCRIPTION:
Anomalies include, but are not limited to:

Posterior Capsule Opacification (PCO) (pathological condition) - delayed clouding of the lens capsule after cataract surgery.

Glistenings - fluid-filled micro-vacuoles that form within the intraocular lens (IOL) optic when the IOL is in an aqueous environment. They may appear to be on the lens surface.

Artifacts - glares, halos, starbursts and/or shadows caused by IOLs.

Fibrosis - the formation of fibrous connective tissue, as in a scar.

Glare - undesirable sensation produced by brightness that is much greater than that to which the eyes are adapted. Causes annoyance, discomfort, or loss in visual performance.

Halos (symptom) - the appearance of hazy ring(s) around light.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the EC-3 clinical trial
* Subjects who were implanted with EC-3 IOL

Exclusion Criteria:

* Removal of the EC-3 IOL at any time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were enrolled in the EC-3 study and implanted with the EC-3 IOL.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the presence, if any, of PCO (Posterior Capsule Opacification) in the EC-3 lens. | 2-3 years post-implantation
  Routine eye exam by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: P. Dee G. Stephenson, M.D., Principal Investigator — Stephenson Eye Associates; N. Timothy Peters, M.D., Principal Investigator — Eyesight Ophthalmic Services PA; Christophe Pey, M.D., Principal Investigator — Cabinet d'Ophtalmologie du Dr. Pey
Locations (3):
- United States (2):
  - Stephenson Eye Associates, Venice, Florida
  - Eyesight Ophthalmic Services, Dover, New Hampshire
- Cabinet d'Ophtalmologie du Dr. Pey, Le Puy-en-Velay, France